CLINICAL TRIAL: NCT03322709
Title: Minimally Invasive Kidney Transplantation: Surgical Stress and Kidney Injury
Brief Title: Minimally Invasive Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 184202
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Transplant;Failure,Kidney
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic-assisted kidney transplant: Adult patients undergoing robotic kidney transplantation. The transplant operation will be undertaken using the da Vinci systems robot in minimally invasive fashion.
  Interventions: Procedure: kidney transplant
- Open kidney transplant: Adult patients undergoing kidney transplantation via an open approach.
  Interventions: Procedure: kidney transplant
- Donor nephrectomy: Adult patients undergoing donor nephrectomy will have a scan of their abdominal wound to compare wound healing.

INTERVENTIONS:
Procedure: kidney transplant — Transplantation of a kidney either by open surgery or robotic assisted laparoscopic surgery.
  Groups: Open kidney transplant; Robotic-assisted kidney transplant

SUMMARY:
This study aims to investigate the effect of robot-assisted laparoscopic kidney transplantation on kidney injury by measuring biomarkers of kidney injury which are found in blood and urine to establish if there is a significant difference between robotic and open surgery. The study will also investigate the potential benefits of minimally invasive surgery on the surgical trauma associated with open surgery by assessing the surgical stress response between groups of kidney transplant patients receiving either open or minimally invasive kidney transplants and by comparing wound healing with patients undergoing donor nephrectomy.

DETAILED DESCRIPTION:
1. Introduction

1.1 Background

Living donor kidney transplantation is the optimal treatment for end stage renal disease (ESKD). This process involves a mandatory period of warm and cold ischaemia before the donor kidney is reperfused. The reperfusion injury causes damage to the transplanted kidney that may affect its long term outcome. In living donor kidney transplantation this period of ischaemia is kept to a minimum. However, minimally invasive kidney transplantation (MIKT) has been shown to increase the warm ischaemia time for these patients due to the prolonged anastomosis time and the graft and patient are exposed to pneumoperitoneum for a significant amount of time. It is not clear if these events affect graft outcomes.

Biomarkers of acute kidney injury are of interest in transplantation as they may be used to assess the severity of graft injury and predict the likely clinical outcomes at an early stage. There is evidence that they can predict delayed graft function after kidney transplantation.

MIKT also has the potential in reducing the surgical trauma associated with open surgery due to smaller incisions; this may reduce infections and improve wound healing. Evidence from laparoscopic donor nephrectomy shows clear benefits to patients.

1.2 Rationale

A key issue arising from MIKT is its effect on the kidney allograft. The robotic kidney transplant technique prolongs the re-warming time due to the longer anastomosis time. Results suggest that this may reduce the glomerular filtration rate (eGFR) in the early post-transplant period when compared to open kidney transplant with no difference in function at 1 and 2 year follow-up. The long-term consequences for the graft beyond this period are unknown. The effects of pneumoperitoneum on the transplant kidney have also been questioned with suggestions that higher intra-abdominal pressures may reduce allograft perfusion during surgery with negative consequences for the allograft based on experience with other studies of both human and animal models. There is unpublished data that suggests that the effects on longer term graft outcomes are not significant.

MIKT promises to offer significant benefits to kidney transplant recipients including less manipulation of the graft during surgery and a reduction in surgical site infections which has already been noted in obese patients undergoing robotic MIKT. Smaller incisions with reduced analgesia requirement are a key benefit which may affect length of stay and associated co-morbidity, hospital costs and the patient experience which has been demonstrated with the donor nephrectomy operation.

The expression of several biomarkers of kidney injury has been demonstrated to reflect damage to the graft and subsequent kidney function in living donor kidney transplantation. These biomarkers, including Kidney Injury Molecule 1 (KIM-1), neutrophil gelatinase associated lipocalin (NGAL) and interleukin 18 (IL-18) are expressed in both serum and urine. Changes in their expression can predict some outcomes after transplantation. These biomarkers offer an advantage over traditional means of assessing kidney injury and function after transplantation such as serum creatinine measurement, urine output and kidney biopsy in that they can be detected early in the spectrum of acute kidney injury.

Patients with ESRD usually have multiple co-morbidities and are less able to withstand the stress of major surgery compared to other patients leading to greater mortality and complications. MIKT may reduce the surgical stress burden for these patients, compared with open surgery, but this is currently uncertain. Evidence from other fields of surgery has shown that the changes in the metabolic stress response to open and minimally invasive surgery can be quantified.

We therefore propose to perform this study to assess the impact of minimally invasive kidney transplantation on the transplant kidney and the recipient by observing the expression of biomarkers and establishing their relationship to outcomes after transplantation.

2 Study Objectives, Design and Statistics 2.1. Study Objectives

This study aims to investigate the effect of the warm ischaemia time and pneumoperitoneum on kidney injury by measuring biomarkers of acute kidney injury which are found in blood and urine to establish if there is a significant difference between robotic and open surgery. The study will also investigate the potential benefits of minimally invasive surgery on the surgical trauma associated with open surgery by assessing the surgical stress response and wound healing between groups of kidney transplant patients receiving either open or minimally invasive kidney transplants. Wound healing will also be compared with patients undergoing a different minimally invasive surgical technique (laparoscopic donor nephrectomy) as they will have a similar incision.

The primary outcome measure is the difference in expression of plasma and serum biomarkers of kidney injury and surgical stress in the recipient groups. The secondary outcomes will include clinical outcomes such as infection, graft function and acute rejection, evidence of wound healing as assessed by ultrasound scan and quality of life outcomes assessed by questionnaire.

2.2 Study Design & Flowchart The study will be conducted on an observational case-control basis comparing groups of patients receiving standard care in three arms: open living donor kidney transplantation, robotic living donor kidney transplantation and laparscopic donor nephrectomy. Biomarkers of kidney injury and the surgical stress response will be measured in plasma and urine of the recipients only.

Participants will receive information leaflets during education sessions prior to transplantation or donor surgery. Information about the study will be given during this period and they will also be approached in clinic prior to surgery to gain their informed consent after they have had the time to consider the information about the study.

Participants will have blood samples collected for the study at the same time as their routine clinical samples are taken wherever possible. These samples will be collected on the day of surgery and all post-operative days until day seven after surgery if they are inpatients. Additional samples will be collected at non-routine times in the first 24 hours after transplant surgery only.

Urine samples will be collected from the catheter during surgery and each post-operative day up till day seven after surgery if they are inpatients.

All participants will be offered the opportunity of undergoing an optional bedside ultrasound scan of their abdominal wall incision at day three post-surgery.

Final blood and urine samples will be collected at the time of the participant's routine post-operative visit at 1 month.

Biomarkers will be measured using Luminex and ELISA techniques as appropriate. The biomarkers to be measured will include Kidney injury molecule 1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL) and Interleukin-18 (IL-18).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years recieving a living donor kidney transplant at our institution

Exclusion Criteria:

* refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal failure patients and donors
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Expression of biomarkers of kidney injury | 30 days post op
  KIM-1, NGAL and Interleukin 18 will be measured pre-op and post operatively up to day 30.

SECONDARY OUTCOMES:
Wound healing | 3 time points post op up to 14 days.
  Assessed by clinical markers such as infection and by ultrasound scan of incisions.

CONTACTS AND LOCATIONS:
Overall Officials: Nizam Mamode, Study Chair — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No